CLINICAL TRIAL: NCT05505968
Title: Evaluation of the Interest of a Virtual Reality Headset on Pain and Anxiety During Epidural Injection Through the Sacrococcygeal Hiatus in Patients With Lumbar Radicular Pain.
Brief Title: Interest of Virtual Reality Headset During Injection in Patients With Back Pain and Sciatica
Acronym: Epi-RéV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PO22085*
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2024-01

CONDITIONS: Lumbar Radicular Pain
MeSH Terms: interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality - Day1 (Experimental): Use of the virtual reality headset during the first epidural infiltration (Day 1). The second infiltration (Day 3) will be performed without the virtual reality headset.
  Interventions: Other: Virtual Reality Headset
- virtual reality - Day3 (Experimental): First epidural infiltration without the virtual reality headset (day 1). The second infiltration will be performed with the virtual reality headset (Day 3).
  Interventions: Other: Virtual Reality Headset

INTERVENTIONS:
Other: Virtual Reality Headset — Virtual Reality Headset of the society Healthy Mind and is a CE Class 1 medical device. This virtual reality headset is a Pico G2 4K and corresponds to the model A7510 and is connected to a Bose Sound Link 2 AE headset.
  Other Names: Medical device

SUMMARY:
For a few years, publications have been published concerning the use of virtual reality headsets in the field of medicine and particularly in various specialities.

It has been evaluated in different studies on pain and anxiety in various medical situations.

A study has shown a correlation between a decrease in pain in a clinical way during a painful stimulation and a decrease in certain areas of the brain.

In this context, the use of the virtual reality headset could then be used in medical interventions that may be painful for the patient.

The lumbar radicular pain is a common disease in the world. The epidural injection is one of the treatment of this pathology. He may be performed to reduce the pain but sometimes this act is painful. Most of the time this procedure is performed without premedication.

To the knowledge of the investigators, there are currently no studies on the assessment of pain under a virtual reality headset during the performance of an epidural injection in rheumatology.

The aim of the study is to demonstrate that the Virtual Reality Headset can reduce the pain and the anxiety during an epidural injection.

DETAILED DESCRIPTION:
Any patient who meets the inclusion criteria can be offered this study. The physician will verify with the data collected during the usual management of the patient whether the patient presents the inclusion criteria and no exclusion criteria. The questioning (history of the disease, treatments, etc.) and the clinical examination will be carried out within the framework of the usual management of the patient before his inclusion in the study.

After the patient's agreement and signature of the consent form, the patient will be randomized in one of the two groups :

* Group 1: Use of the virtual reality headset during the first epidural infiltration. The second infiltration will be performed without the virtual reality headset.
* Group 2: First epidural infiltration without the virtual reality headset. The second infiltration will be performed with the virtual reality headset.

The duration of participation in each of the two groups is 3 days:

- On the 1st day, the patients will have to fill in a questionnaire with socio-demographic data, pain related to the disease, their anxiety in general life, their anxiety before the infiltration.

The patient will choose, with the help of the doctor, the landscape that will be projected in the virtual reality headset, and then the helmet will be put in place, again with the help of the doctor.

Concerning the installation, the patient will be in prone position with the hands under the chin with the reality headset so that he cannot rest on the bed. The patient must be comfortable.

The first epidural infiltration will be performed with or without the virtual reality headset depending on the randomization group.

Then the patient will have to estimate his pain thanks to the numerical scale as well as his state of anxiety during the procedure. This part of the questionnaire will be completed after the first infiltration.

* On the 2nd day, there will be no infiltration and no questionnaire to fill in.
* On the 3rd day, the second epidural infiltration will be performed with or without virtual reality headset depending on the randomization group. Patients will be asked to fill in their anxiety status before the procedure, their pain during the procedure and the estimated anxiety during the procedure.

Both infiltrations will be performed by a person trained and experienced in performing infiltrations through the hiatus route.

The virtual reality headset used is provided by the company Healthy Mind and corresponds to a class 1 CE medical device. This virtual reality headset is a Pico G2 4K and corresponds to the model A7510 and is connected to a Bose Sound Link 2 AE headset, all connected to a tablet allowing to control the chosen universe.

There will be no remote monitoring of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18-90 years,
* Diagnosed with lomboradiculalgia requiring two epidural injection through the sacrococcygeal hiatus,
* Hospitalized in the Rheumatology Department of the University Hospital of Reims,
* Speak French language.
* Affiliated or beneficiary of a social security scheme
* Having given their written agreement to participate in the study (signature of the consent form)

Exclusion Criteria:

* Profound or total deafness,
* Visually impaired,
* Presence of contraindication to injection,
* Inability to answer the questionnaire due to severe cognitive impairment,
* Injection with and without virtual reality headset not performed by the same person,
* Vestibular pathologies,
* Epilepsy,
* Claustrophobia,
* Use of nitrous oxide for injection.
* Premedication for infiltration (analgesic, anxiolytic)
* Patients under guardianship, curatorship, safeguard of justice
* Pregnant women
* Psychotic disorders

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory | Day 1
  State-Trait Anxiety Inventory STAI-B (trait anxiety), STAI-A (state anxiety)
State-Trait Anxiety Inventory | Day 3
  STAI-B (trait anxiety), STAI-A (state anxiety)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Result] Javelot M, Chopin C, Bolko L, Hittinger A, Geoffroy M, Charlot I, Adeline F, Coutureau C, Duvivier A, Salmon JH. Effect of Virtual Reality on Pain and Anxiety During Epidural Steroid Injection in Patients with Lumbar Radicular Pain: An Open-Label Randomized Trial. Healthcare (Basel). 2025 Sep 22;13(18):2376. doi: 10.3390/healthcare13182376. PMID 41008506